CLINICAL TRIAL: NCT00520013
Title: A Randomized Phase II Trial of Avastin (A) or Avastin and Erlotinib (AE) as First Line Consolidation Chemotherapy After Carboplatin, Paclitaxel, and Avastin (CTA) Induction Therapy for Newly Diagnosed Advanced Ovarian, Fallopian Tube, Primary Peritoneal Cancer & Papillary Serous or Clear Cell Mullerian Tumors
Brief Title: Avastin +/- Erlotinib Consolidation Chemotherapy After Carboplatin, Paclitaxel, and Avastin (CTA) Induction Therapy for Advanced Ovarian, Fallopian Tube, Primary Peritoneal Cancer & Papillary Serous or Clear Cell Mullerian Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susana M. Campos, MD, Medical Oncologist., Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-039
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Papillary Serous Mullerian Tumor; Clear Cell Mullerian Tumor
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- carboplatin/paclitaxel/bevacizumab then bevacizumab (Experimental): Induction (CTA): Patients received carboplatin IV AUC 5, paclitaxel IV 175 mg/m2 and bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle for 6 cycles. Bevacizumab started with cycle 2.
  Patients with disease progression based on radiographic evaluation after induction could not advance to the randomized consolidation phase.
  Consolidation (A): Patients received bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle for 1 year.
  Interventions: Drug: bevacizumab; Drug: paclitaxel; Drug: carboplatin
- carboplatin/paclitaxel/bevacizumab then bevacizumab/erlotinib (Experimental): Induction (CTA): Patients received carboplatin IV AUC 5, paclitaxel IV 175 mg/m2 and bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle for 6 cycles. Bevacizumab started with cycle 2.
  Patients with disease progression based on radiographic evaluation after induction could not advance to the randomized consolidation phase.
  Consolidation (AE): Patients received bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle and oral erlotinib 150mg daily for 1 year.
  Interventions: Drug: bevacizumab; Drug: erlotinib; Drug: paclitaxel; Drug: carboplatin
- carboplatin/paclitaxel/bevacizumab (Experimental): Induction (CTA): Patients received carboplatin IV AUC 5, paclitaxel IV 175 mg/m2 and bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle for 6 cycles. Bevacizumab started with cycle 2.
  Patients with disease progression based on radiographic evaluation after induction could not advance to the randomized consolidation phase.
  Consolidation: None
  Interventions: Drug: bevacizumab; Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: bevacizumab
  Other Names: Avastin; rhuMAB VEGF
Drug: erlotinib
  Other Names: Tarceeva
  Arms: carboplatin/paclitaxel/bevacizumab then bevacizumab/erlotinib
Drug: paclitaxel
  Other Names: Taxol
Drug: carboplatin
  Other Names: Paraplatin

SUMMARY:
The purpose of this research study is to evaluate how patients with newly diagnosed advanced ovarian, fallopian tube, primary peritoneal cancer and papillary serous or clear cell mullerian tumors respond to consolidation therapy with Avastin and erlotinib or Avastin alone over 1 year. These drugs have been used in the treatment of other types of cancers and information from those studies suggests that these agents may help to treat the cancers studied here.

DETAILED DESCRIPTION:
Objectives:

Primary To examine the progression free survival (PFS) of Avastin and Erlotinib (AE) or Avastin (A) as consolidation therapy.

Secondary To examine the toxicity between the two consolidative regimens AE vs. A. To assess the response rate of CTA.

STATISTICAL DESIGN This study uses a randomized selection design. Both consolidation treatment arms are deemed experimental and are compared against a historical control [McGuire WP et al. Cyclophosphamide and cisplatin compared with paclitaxel and cisplatin in patients with stage III and stage IV ovarian cancer. NEJM 1996: 334:1-6. PMID:7494563]. With 30 patients in a given arm and 6 months of follow-up, there was 80% power to detect a 61.5% increase in median PFS from 13 months to 21 months assuming 1-sided 10% significance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Histological diagnosis of epithelial ovarian carcinoma, fallopian tube cancer, primary peritoneal carcinoma, or papillary serous mullerian carcinoma
* Previous attempted surgical debulking
* Stage III or IV
* Willing and able to undergo second look laparoscopy
* Performance status 0-1 by ECOG scale
* Peripheral neuropathy < grade 2
* Life expectancy of 6 months or greater

Exclusion Criteria:

* Patients with clinically significant cardiovascular disease as outlined in the protocol
* Neutrophil count < 1,500/mm3; platelet count <100,000/m3
* Alkaline phosphatase or bilirubin > 1.5 x ULN, SGOT > 5 x ULN
* Calculated creatinine clearance < 50ml/min
* Prior chemotherapy or radiotherapy for other malignancy except for the treatment for localized breast cancer greater than five years prior to diagnosis
* No more than one cycle of first line chemotherapy with carboplatin and paclitaxel
* Inadequate surgical cytoreduction such that interval cytoreductive surgery could materially improve prognosis
* Concurrent invasive malignancy
* Evidence of bleeding diathesis or coagulopathy
* Evidence of tumor involving major blood vessels on any prior CT scans
* Surgical wound that has failed to close
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of this study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 0
* Serious non-healing wound, ulcer, or bone fracture
* Prior treatment with an anti-angiogenic agent
* Any active bleeding
* Active psychiatric disease or neurologic symptoms requiring treatment
* Presence of central nervous system brain metastases
* Proteinuria at screening as demonstrated by criteria in protocol
* Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent
* Known hypersensitivity to Cremophor EL or any component of Avastin
* Active bacterial, viral, or fungal infections
* Receiving any other investigational agent
* History of gastrointestinal perforation
* Prior therapies targeting the epidermal growth factor receptor
* Symptoms of bowel obstruction
* Dependence on TPN or IV hydration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Campos, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty patients were enrolled between Aug 3, 2007 and Jan 6, 2010.
Pre-assignment Details: Patients with disease progression based on radiographic evaluation after induction could not advance to the randomized consolidation phase.
Period: Overall Study
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib | Carboplatin/Paclitaxel/Bevacizumab
Started | 23 | 25 | 11 (Excludes a pt who went off-study (on reg day) due to consent that may not have been informed (ESL).)
Treated | 23 | 25 | 11
Completed | 11 | 10 | 0
Not Completed | 12 | 15 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 2 | 10 | 7
Not completed — Progressive Disease | 7 | 3 | 0
Not completed — Clinical Progression | 3 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of treated patients.
Groups:
- Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab: Induction (CTA): Patients received carboplatin IV AUC 5, paclitaxel IV 175 mg/m2 and bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle for 6 cycles. Bevacizumab started with cycle 2.
  Patients with disease progression based on radiographic evaluation after induction could not advance to the randomized consolidation phase.
  Consolidation (A): Patients received bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle for 1 year.
  bevacizumab
  paclitaxel
  carboplatin
- Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib: Induction (CTA): Patients received carboplatin IV AUC 5, paclitaxel IV 175 mg/m2 and bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle for 6 cycles. Bevacizumab started with cycle 2.
  Patients with disease progression based on radiographic evaluation after induction could not advance to the randomized consolidation phase.
  Consolidation (AE): Patients received bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle and oral erlotinib 150mg daily for 1 year.
  bevacizumab
  erlotinib
  paclitaxel
  carboplatin
- Carboplatin/Paclitaxel/Bevacizumab: Induction (CTA): Patients received carboplatin IV AUC 5, paclitaxel IV 175 mg/m2 and bevacizumab IV 15 mg/kg on day 1 (+/- 3d) of a 21 day cycle for 6 cycles. Bevacizumab started with cycle 2.
  Patients with disease progression based on radiographic evaluation after induction could not advance to the randomized consolidation phase.
  Consolidation: None
  bevacizumab
  paclitaxel
  carboplatin
- Total: Total of all reporting groups
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib | Carboplatin/Paclitaxel/Bevacizumab | Total
Number analyzed (Participants) | 23 | 25 | 11 | 59
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [48 to 63] | 56 [49 to 61] | 54 [51 to 59] | 57 [49 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 11 | 59
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 11 | 59
Cancer Type [Number; unit: participants]
  Primary peritoneal | 4 | 1 | 1 | 6
  Fallopian tube | 5 | 4 | 1 | 10
  Epithelial ovarian | 10 | 17 | 8 | 35
  Uterine papillary serous | 2 | 1 | 1 | 4
  Other (mixed, carcinosarcoma) | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Consolidation Progression-Free Survival
Description: Consolidation PFS based on the Kaplan-Meier method was defined as the time from the first day of consolidation therapy to documented disease progression (PD) or disease-specific death. Based on RECIST 1.1, radiographic PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum since beginning consolidation, the appearence of one or more new lesions and/or unequivocal progression of existing non-target lesions. Based on Rustin criteria, serlogic PD was a rise in CA125 since beginning of consolidation or previously normal CA125 that rises to >/= 2xULN with either event documented on 2 occasions. Patients who were event-free were censored at the date of their last disease evaluation.
Time Frame: Assessments occurred every cycle (serologic) and every 3 cycles (radiologic) on consolidation treatment. Pts were allowed on consolidation therapy for up to 1 year and upon treatment discontinuation were followed for another year.
Population: The analysis dataset is comprised of patients randomized to consolidation treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib
Number analyzed (Participants) | 23 | 25
months | 13.3 [10.1 to NA] — PFS data was not mature enough to provide an upper bound on 95% CI. Also note per design each arm was separately compared to a historical control [PMID:7494563]. | 18.9 [15.4 to NA] — PFS data was not mature enough to provide an upper bound on 95% CI. Also note per design each arm was separately compared to a historical control [PMID:7494563].

2. Primary Outcome: Consolidation Treatment-related Toxicity Rate
Description: Consolidation treatment-related toxicity rates based on CTCAEv3 were defined as rates of maximum grade 3 or higher toxicity events with attribution possible, probable or definite occurring during consolidation treatment and up to 30 days post-treatment.
Time Frame: Assessed every cycle during consolidation treatment and up to 30 days post-treatment. Per protocol, consolidation treatment was a fixed duration of 1 year.
Population: The analysis dataset is comprised of patients who were randomized to consolidation treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib
Number analyzed (Participants) | 23 | 25
percentage of participants | 30.4 [13.2 to 52.9] | 72.0 [50.6 to 88.0]

3. Secondary Outcome: Consolidation Objective Response Rate
Description: Consolidation objective response (OR) was based on RECIST 1.0 criteria with OR defined as achieving partial response (PR) or complete response (CR). Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. For CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. If CA125 disease then OR based on Rustin criteria is a 50% decrease in serum CA125 level from two initially elevated samples confirmed by a 4th sample.
Time Frame: Assessments occurred every cycle (serologic) and every 3 cycles (radiologic) on consolidation treatment. Pts were allowed on consolidation therapy for up to 1 year.
Population: The analysis dataset is comprised of all patient who started consolidation treatment.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib
Number analyzed (Participants) | 23 | 25
proportion of patients | 0.65 [.43 to .84] | .60 [.39 to .79]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout consolidation treatment from time of first dose and up to day 30 post-treatment. Per protocol, consolidation treatment was a fixed duration of 1 year.
Description: Serious and other AE data is only available for consolidation treatment reflecting the primary and secondary study objectives centered on the evaluation of consolidative regimens AE vs A.
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib
Serious Adverse Events (participants affected / at risk) | 7/23 | 18/25
Other Adverse Events (participants affected / at risk) | 23/23 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab (N=23) | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib (N=25)
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 5
Enteritis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Infection-other (Infections and infestations) | 0 | 1
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Irregular menses (Reproductive system and breast disorders) | 0 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 6 | 4
Hemorrhage-other (Vascular disorders) | 0 | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab (N=23) | Carboplatin/Paclitaxel/Bevacizumab Then Bevacizumab/Erlotinib (N=25)
Abdomen, pain (Gastrointestinal disorders) | 3 | 1
Alkaline phosphatase (Investigations) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 11
ALT, SGPT (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 5
Anxiety (Psychiatric disorders) | 5 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
AST, SGOT (Investigations) | 0 | 2
Bicarbonate (Metabolism and nutrition disorders) | 1 | 0
Bilirubin (Investigations) | 0 | 1
Bladder, pain (Renal and urinary disorders) | 0 | 1
Bone, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 0 | 1
Chest/thoracic pain NOS (General disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 6
Constitutional, other (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
C-P arrest, non-fatal, cause unk (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dental/teeth/peridontal (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5 | 18
Dizziness (Nervous system disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 11
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Edema limb (General disorders) | 1 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Face, pain (General disorders) | 1 | 0
Fatigue (General disorders) | 18 | 21
Fever w/o neutropenia (General disorders) | 0 | 2
GI-other (Gastrointestinal disorders) | 0 | 3
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Head/headache (Nervous system disorders) | 6 | 4
Hemoglobin (Blood and lymphatic system disorders) | 8 | 8
Hemorrhage-other (Vascular disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 9 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 8
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3
Hypotension (Vascular disorders) | 0 | 1
Infection Gr0-2 neut, lip/perioral (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, meninges (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1 | 1
Infection Gr0-2 neut, wound (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, anal/perianal (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, skin (Infections and infestations) | 0 | 1
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 0 | 2
Infection-other (Infections and infestations) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Intestine, pain (Gastrointestinal disorders) | 1 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 12 | 7
Joint-function (Musculoskeletal and connective tissue disorders) | 0 | 3
Leukocytes (Investigations) | 3 | 5
Libido (Psychiatric disorders) | 0 | 1
Lip, pain (Gastrointestinal disorders) | 0 | 1
Lymphatics-other (Blood and lymphatic system disorders) | 0 | 1
Metabolic/Laboratory-other (Investigations) | 0 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 4
Muco/stomatitis (symptom) stomach (Gastrointestinal disorders) | 0 | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 0 | 2
Muscle, pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 | 2
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 5 | 9
Neck, pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neurologic-other (Nervous system disorders) | 1 | 0
Neuropathy-motor (Nervous system disorders) | 2 | 3
Neuropathy-sensory (Nervous system disorders) | 14 | 12
Neutrophils (Investigations) | 1 | 5
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Nonneuropathic upper extr muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 2
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 13 | 7
Oral cavity, hemorrhage (Gastrointestinal disorders) | 3 | 1
Oral cavity, pain (Gastrointestinal disorders) | 0 | 3
Oral gums, pain (Gastrointestinal disorders) | 1 | 0
Pain-other (General disorders) | 2 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Platelets (Investigations) | 5 | 1
Proteinuria (Renal and urinary disorders) | 4 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 5
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 8
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 16
Rectum, hemorrhage (Gastrointestinal disorders) | 1 | 0
Renal/GU-other (Renal and urinary disorders) | 1 | 1
Rigors/chills (General disorders) | 0 | 2
Salivary (Gastrointestinal disorders) | 0 | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin, pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 4
Sinus, pain (Nervous system disorders) | 1 | 0
Taste disturbance (Nervous system disorders) | 1 | 3
Throat/pharynx/larynax, pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 1
Urinary hemorrhage NOS (Renal and urinary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vagina, hemorrhage (Reproductive system and breast disorders) | 2 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Vision-blurred (Eye disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Weight loss (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No